CLINICAL TRIAL: NCT05219786
Title: Online Field Test of an Appendicitis Decision Support Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, David Flum, Professor of Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00012210
Record Dates: First submitted 2021-11-08; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Appendicitis Acute
Keywords: decision support; decision aid; decisional conflict
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Support Tool (Experimental): In this arm study participants saw a decision support tool consisting of a video and a interactive decision aid (www.appyornot.org).
  Interventions: Behavioral: Appendicitis Decision Support Tool
- Infographic (Active Comparator): Participant saw a static infographic providing information about the two treatments for appendicitis.
  Interventions: Behavioral: Control Infographic

INTERVENTIONS:
Behavioral: Appendicitis Decision Support Tool — Viewing of a decision support tool.
  Arms: Decision Support Tool
Behavioral: Control Infographic — Viewing of a standardized infographic
  Arms: Infographic

SUMMARY:
After the recent publication of the CODA Trial comparing antibiotics and surgery for acute appendicitis, the investigators developed a comprehensive decision support tool. This tool will help patients understand the risks and benefits of each treatment and make a treatment decision. This study is an online randomized field test comparing the decision support tool to a control infographic and assessing it's affect on decisional outcomes, such as decisional conflict.

ELIGIBILITY:
Inclusion Criteria: who live in the United States and who have not previously had appendicitis.

* Workers on Amazons Mechanical Turk Platform with an approval rating of 95% or higher
* Workers on Amazons Mechanical Turk Platform who live in the United States
* Workers on Amazons Mechanical Turn Platform who have not previously had appendicitis

Exclusion Criteria:

* Employees or relatives of employees of the University of Washington

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Pre vs. Post Intervention | At time of enrollment
  Assessed using the validated decisional conflict scale comparing only participants in the intervention arm before and after viewing the decision support tool.

SECONDARY OUTCOMES:
Decisional Conflict Between Arms | At time of enrollment
  Total score on the validated decisional conflict scale after viewing the intervention support tool or the control infographic. Scale ranges from 0-100 with higher scores being worse.
Acceptability | At time of enrollment
  Between arm comparison of the acceptability of the information presented to the participants rated on a 4 point acceptability scale with higher scores representing higher acceptability.
Trust and Accuracy of Information | At time of enrollment
  Participants perception of the trustworthiness and accuracy of the information presented to them on a 5 point scale with higher scores representing a higher perceived trustworthiness and perceived accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] CODA Collaborative; Flum DR, Davidson GH, Monsell SE, Shapiro NI, Odom SR, Sanchez SE, Drake FT, Fischkoff K, Johnson J, Patton JH, Evans H, Cuschieri J, Sabbatini AK, Faine BA, Skeete DA, Liang MK, Sohn V, McGrane K, Kutcher ME, Chung B, Carter DW, Ayoung-Chee P, Chiang W, Rushing A, Steinberg S, Foster CS, Schaetzel SM, Price TP, Mandell KA, Ferrigno L, Salzberg M, DeUgarte DA, Kaji AH, Moran GJ, Saltzman D, Alam HB, Park PK, Kao LS, Thompson CM, Self WH, Yu JT, Wiebusch A, Winchell RJ, Clark S, Krishnadasan A, Fannon E, Lavallee DC, Comstock BA, Bizzell B, Heagerty PJ, Kessler LG, Talan DA. A Randomized Trial Comparing Antibiotics with Appendectomy for Appendicitis. N Engl J Med. 2020 Nov 12;383(20):1907-1919. doi: 10.1056/NEJMoa2014320. Epub 2020 Oct 5. PMID 33017106
- See also: Decision Support Tool — http://www.appyornot.org